CLINICAL TRIAL: NCT04511182
Title: Early Individualized-exercise Based Cardiac Rehabilitation Program in Patients With a Recent Acute Myocardial Infarction (EARLYmyo-CRPⅡ): Study Protocol for a Randomised Controlled Trial
Brief Title: Early Individualized-Exercise Based Cardiac Rehabilitation Programs in Patients With Acute Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRP2
Record Dates: First submitted 2020-08-05; First posted 2020-08-13 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise intervention group (Experimental): Patients will receive standard medications plus EBCR 。Education covering topics related to AMI and exercise for AMI will be implemented and any consultations on exercise prescription and disease management will be explained by a cardiac rehabilitation team consisting of cardiologists, cardiology nurses and physiotherapists.
  Interventions: Behavioral: Exercise-based cardiac rehabilitation
- Usual care group（control） (No Intervention): Patients will receive standard medications according to national guidelines, as well as education and consultations as intervention group. However，no exercise prescription is given,

INTERVENTIONS:
Behavioral: Exercise-based cardiac rehabilitation — Exercise program is based on aerobic exercise and supplemented by strength training following the principle of gradual improvement. The type of exercise, such as walking, jogging, cycling, and the intensity of exercise which is recommended to use a cardiotach or pedometer to detect, are both defined by the results of CPET, such as METs value. Participators must be prepared for about 5-10 minutes to warm up and recover before and after exercise. 30-50 minutes a day, 5 days a week, with a total exercise time of not less than 150 minutes per week. It can be carried out in different stages according to the physical condition. After 1-3 months, the exercise prescription will be re-adjusted according to the results of reexamination.
  All patients will undergo Cardiopulmonary Exercise Test, SF-36, echocardiography and laboratory examination prior to initiation of the trial, and which will be checked again after 3 months, and 6 months.
  Arms: exercise intervention group

SUMMARY:
Acute myocardial infarction (AMI) is a life-threatening condition and a cause of functional disability. After reperfusion therapies and pharmacological strategies, patients suffered great pain physically and mentally. How to improve the quality of life and the prognosis in patients with AMI is a hot topic in the field of cardiac rehabilitation now. In this study, a randomized, controlled and prospective clinical trial is designed for patients with AMI to improve exercise capacity, cardiometabolic parameters, as well as quality of life by an individualized, low-cost exercise intervention we developed after evaluation by Cardiopulmonary Exercise Tests (CPET). Serial CPET are performed to prospectively measure changes in aerobic exercise capacity, and the MOS item short form health survey（SF-36）are constructed to survey life quality. What's more, echocardiography and NT-proBNP are also assessed.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a life-threatening condition and a cause of functional disability, although reperfusion therapies and pharmacological strategies have been developed dramatically. Percutaneous coronary intervention（PCI）can effectively improve the myocardial blood supply of patients, However, various degrees of reduced exercise tolerance, anxiety and depression symptoms, impaired social function may occur after PCI and then lead to the decline of their quality of life. Exercise-based cardiopulmonary rehabilitation, which has beneficial effects on physical fitness, quality of life, cardiovascular risk factors and clinical outcome, is an important part of secondary prevention for patients after an acute myocardial infarction. Despite the evidence of these beneficial effects, cardiac rehabilitation programs are still largely underutilized and the exact benefits are still less well known. In this study, a randomized, controlled and prospective clinical trial is designed for patients with AMI to improve exercise capacity, cardiometabolic parameters, as well as quality of life by an individualized, low-cost exercise intervention we developed after evaluation by Cardiopulmonary Exercise Tests (CPET) . Serial CPET are performed to prospectively measure changes in aerobic exercise capacity, and the MOS item short form health survey（SF-36）are constructed to survey life quality. What's more, echocardiography and NT-proBNP are also assessed.

ELIGIBILITY:
Inclusion criteria

1. Acute myocardial infarction (AMI) within 1 months prior to recruitment.
2. Complete revascularization.
3. Man or non- pregnant women aged from 18 to 80 years.

Exclusion criteria

1. Uncontrolled hypertension (systolic blood pressure/diastolic blood pressure >160/100 mmHg)，or symptomatic hypotension.
2. Significant resting electrocardiogram abnormalities (left bundle branch block, non-specific intraventricular conduction delay, left ventricular hypertrophy, resting ST-segment depression), life-threatening cardiac arrhythmias.
3. Acute myocarditis, pericarditis or acute systemic illness.
4. Those who are assessed by the doctor as high-risk [12].
5. Pacemaker or implantable cardioverter defibrillator.
6. Any contraindication to exercise testing or exercise training or inability to complete a CPET.
7. Life-threatening diseases with limited life expectancy <3 year.
8. Uncontrolled unstable angina pectoris.
9. Significant valvular disease (mitral stenosis, moderate to severe mitral insufficiency, aortic stenosis, or aortic insufficiency, severe mitral / aortic regurgitation).
10. Severe mental or cognitive impairment.
11. Inability to follow the procedures of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2)change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in peak VO2 comparing Experimental group with control.

SECONDARY OUTCOMES:
Ventilatory efficiency (VE/VCO2 slope) change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in Ventilatory efficiency (VE/VCO2 slope) comparing experimental group with control.
oxygen consumption (VO2) at anaerobic threshold | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in VO2 at anaerobic threshold comparing Experimental group with control.
Oxygen uptake related to work rate（ΔVO2/ΔWR）change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in Oeygen uptake related to work rate（ΔVO2/ΔWR）comparing experimental group with control.
Peak /AT Oxygen Pulse (O2-Pulse)change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in Peak /AT Oxygen Pulse (O2-Pulse) comparing experimental group with control.
Peak metabolic equivalent (MET) change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in peak metabolic equivalent (MET) change comparing experimental group with control.
Heart rate variability | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in Heart rate variability comparing experimental group with control.
Body mass index（BMI）change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in Body mass index（BMI）comparing experimental group with control. BMI is the value obtained by dividing body weight by height square (weight in kilograms, height in meters). BMI is a standard commonly used in the world to measure the degree of obesity and health of the human body.
LVEF change | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in LVEF comparing experimental group with control.
NT-proBNP(pg/ml) | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in NT-proBNP comparing Experimental group with control.
The MOS item short form health survey(SF-36) | Baseline, 3, 6 months
  Difference in the interval changes from baseline to 3 months and 6 months in The MOS item short form health survey(SF-36) comparing experimental group with control.
The occurrence and composite of major adverse cardiac events (MACE) | 3, 6 months
  Major adverse cardiac events (MACE) included all-cause mortality, non-fatal myocardial infarction and coronary revascularisation. we check the outcome in 3 months and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Shao, M.D,Ph.D, Study Chair — RenJi Hospital; Jun Ma, M.D,Ph.D, Study Director — RenJi Hospital
Locations (1):
- RenJi Hospital, Shanghai JiaoTong University, School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No